CLINICAL TRIAL: NCT05322928
Title: Promotion of Physical Activity Through Telehealth-delivered Support of Engagement in Daily Occupations
Brief Title: Physically Active Through Daily Occupations With Telehealth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Slagelse Hospital (Other)
Collaborators: Naestved Hospital (Other)
Responsible Party: Principal Investigator, Svetlana Solgaard Nielsen, Principal Investigator, Slagelse Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSN
Record Dates: First submitted 2022-03-17; First posted 2022-04-12 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Chronic Pain
Keywords: activities of daily living; habits; health behavior; occupational therapy; sedentary lifestyle
MeSH Terms: conditions — Chronic Pain; Habits; Health Behavior; Sedentary Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Engagement in daily occupations (Experimental): The experimental contents will include 1-hour video appointments with an occupational therapist a week in four weeks and a maintenance phase of similar session format every second week in two months.
  Interventions: Behavioral: Engagement in daily occupations

INTERVENTIONS:
Behavioral: Engagement in daily occupations — The 12-week occupational therapy individual person-centered intervention will be delivered by an occupational therapist according to the individual intervention plan, with a 1-hour video appointment (Region Zealand VDX-connection) a week in four weeks and a maintenance phase of similar session format every second week in two months.
  The intervention will include identification of occupational problems that limit compliance with the PA recommendations, setting tailored occupational goals to enhance physically active lifestyle, supervised goal work and goal evaluation. Through active involvement in value-based prioritizing, planning and performance of meaningful everyday activities, the participants will reduce their sedentary time. Changing health behaviour in a stepwise manner, the participants will become prepared for continuous lifestyle goal work as self-management which will allow for sustainable lifestyle changes, and thus, improved long-term health and quality of life.

SUMMARY:
Background: Previous research has demonstrated that people living with chronic pain who were physically active could better protect themselves from chronicity. Chronic pain population has high motivation for initiating lifestyle changes as a part of their multidisciplinary chronic pain treatment but are often not offered any intervention to improve lifestyle.

Objectives: The project will evaluate feasibility of a telehealth-delivered intervention to promote compliance with current WHO recommendations on weekly moderate-to-vigorous physical activity (MVPA) through increased engagement in daily occupations in adults living with chronic. The feasibility evaluation will inform the design and conduct of a future randomised controlled trial (RCT).

Method: Forty adults over 18 years old, living a sedentary lifestyle (i.e., self-reported MVPA<150 min./ week) and completed their standard specialized multidisciplinary chronic pain rehabilitation at Naestved hospital will be invited to participate in this one-group pretest-post-test study. A mixed methods methodology will be applied to investigate in feasibility outcomes (primary) with green-amber-red method, moderate-to-vigorous physical activity, occupational performance and satisfaction and occupational balance in meaningful daily activities, pain spreading, pain intensity, central sensitization, pain self-efficacy, pain catastrophizing, health-related quality of life (HRQoL) and satisfaction with the treatment.

With inspiration from a previous research project with a three-fold focus on meaningful activities, physical activity and eating habits that demonstrated the potential of occupational therapy in lifestyle management in the everyday context, the 12-week occupational therapy individual person-centered intervention will include 1-hour video appointments a week in four weeks and a maintenance phase of similar session format every second week in two months. Individual interviews will add in-depth knowledge on the patients' opinions on the intervention's mechanism and design.

DETAILED DESCRIPTION:
Methods Design A mixed methods feasibility study will be applied to investigate whether MVPA level in adults living with chronic pain can be optimized with an occupational therapy telehealth intervention. One-group pretest-post-test study will assess feasibility outcomes with green-amber-red method, MVPA, occupational performance and satisfaction and occupational balance in meaningful daily activities, pain spreading, pain intensity, central sensitization, pain self-efficacy, pain catastrophizing, health-related quality of life (HRQoL) and satisfaction with the treatment. Individual interviews will add in-depth knowledge on the patients' opinions on the intervention's mechanism and design. The participants' activity diary notes will support the quantitative and qualitative data collected.

Participants The project participants will represent adults living with chronic pain and referred to tertiary chronic pain rehabilitation at a hospital.

Inclusion criteria: Adults over 18 years old, living a sedentary lifestyle (i.e., self-reported MVPA <150 min./ week) and diagnosed with fibromyalgia or musculoskeletal pain in low back, knees, legs, neck, arms and shoulders, who completed their chronic pain treatment at the Multidisciplinary Pain Centre (MPC) at Naestved hospital will be invited to participate.

Exclusion criteria: Adults referred to other specialized treatments or health services (e.g., delivered by rheumatologists, psychiatrists, physiotherapists or multidisciplinary) after the tertiary chronic pain rehabilitation, not sufficient Danish writing and speaking proficiency to allow independent questionnaire completion and translation-free conversation.

Settings Occupational Therapy Unit (OTU) at Naestved hospital in collaboration with the Multidisciplinary Pain Centre (MPC)

Recruitment The MPC team will invite the patients who are discharged from tertiary chronic pain rehabilitation to complete a digital PA survey and will transfer contact information on the patients to the principal investigator (SSN) via Sundhedsplatformen's research list for the project.

The principal investigator will distribute the PA survey to the patients' ID-based secure mail. The principal investigator will invite those who reported MVPA <150 min./ week to participate in an online information meeting about the project (Region Zealand VDX-connection). After considering their participation for one week, the patients who provide informed consent on participation will be included.

Two of the participants will be invited to function as reference persons, to ensure adequate user involvement in the intervention feasibility evaluation and preparation of the RCT. All the participants will be invited to participate in the qualitative interviews after the intervention discharge (Region Zealand VDX connection). A representative sample regarding age, sex and geographical area within Region Zealand will be included for the interviews.

Intervention The 12-week occupational therapy individual person-centered intervention will start from the participants' baseline appointment at the OTU. The experimental contents will be delivered by an occupational therapist according to the individual intervention plan, with a 1-hour video appointment (Region Zealand VDX-connection) a week in four weeks and a maintenance phase of similar session format every second week in two months. After three months in total, the participants will meet for a follow-up assessment and discharge from the intervention.

The intervention is inspired by a previous research project with a three-fold focus on meaningful activities, physical activity and eating habits that demonstrated the potential of occupational therapy in lifestyle management in the everyday context. The intervention will include identification of occupational problems that limit compliance with the PA recommendations, setting tailored occupational goals to enhance physically active lifestyle, supervised goal work and goal evaluation. Through active involvement in value-based prioritizing, planning and performance of meaningful everyday activities, the participants will reduce their sedentary time. Changing health behaviour in a stepwise manner, the participants will become prepared for continuous lifestyle goal work as self-management which will allow for sustainable lifestyle changes, and thus, improved health and quality of life in the long term.

Providers At the start of the project, the intervention will be delivered by the principal investigator who is a graduated occupational therapist with 13 years of experience. Later, additional intervention providers (graduated occupational therapists from the OUT) will be involved.

Assessment The pre-post intervention assessments will take place at the OTU at Naestved Hospital in a quiet room reserved for the purpose. Assessment sessions will not require any specific prerequisites in the participants. Caretakers will be allowed to participate in the assessment sessions. For assessments in paper form, separate files will be used at the baseline and follow-up, to prevent the assessor bias.

Outcomes The choice of the intervention outcomes is guided by the study objectives, The Medical Research Council framework for developing and evaluating complex interventions and the IMMPACT recommendations and include outcomes related to the intervention feasibility, physical health (MVPA time and walking steps), everyday activity (occupational performance and satisfaction, and occupational balance), pain (central sensitization, pain spreading, pain intensity and pain self-efficacy), psychological state (pain catastrophizing), sleep (sleep quality), general well-being (HRQoL) and treatment satisfaction.

Quantitative & quantifiable outcomes A. Feasibility outcomes will be primary outcomes for the project. Feasibility: Feasibility of the procedures planned will be assessed using predefined research progression criteria evaluated by the green-amber-red method. The green-amber-red method where GREEN: Proceed with RCT/implementation; AMBER: Proceed, but changes to the protocol need to be discussed and solved; and RED: Do not proceed unless the problem can be solved, will help evaluate the readiness of the intervention to be tested for effectiveness in an RCT. The predefined research progression criteria will be set for the recruitment; participant retention; program adherence; patients' self-perceived relevance; timing and mode of delivery; assessment procedure acceptance; adverse events; fidelity of delivery; and contextual appropriateness. Detailed description of adverse events is provided below, in a separate section.

B. Secondary outcomes will be assessed before and after intervention.

Qualitative outcomes Individual opinions on the intervention and its self-perceived outcomes will be collected post-intervention. Important themes will be extracted from the transcribed interview data.

Sample size No formal sample size will be calculated. A convenient sample of 30 patients will be included in the project in total, preferably representing different age and sex groups and geographical areas within the Region Zealand. All the participants will be invited to participate in the individual interviews post-discharge. A minimum of 6 patients will be attempted included in the interviews, to ensure data saturation.

Analysis Quantitative analyses: According to the normality check results, the data will be described by mean ± SD or median(range) and analyzed for pre-post changes. Parametric or nonparametric statistics will be applied to the data analysis performed using the STATA 17.0 software (StataCorp, Texas, USA).

Qualitative analysis: The interview data will be transcribed verbatim and analyzed with the thematic analysis methodology.

Results Primary outcomes will inform further research steps and the intervention potential for implementation. Secondary outcomes are expected to improve during the intervention but vary in degree among the participants.

Ethics Digital data will be stored in the project's SharePoint (registration of participation), Redcap database (survey data) and encrypted USB (interview data). Data in paper form will be stored at the OTU at a double-locked location. Access to the project data will be sought granted by a formal agreement from the Data Protection Committee for any person involved in data collection and management.

The project will be approved by the Data Protection Committee of Region Zealand and follow the World Medical Association (WMA) Declaration of Helsinki. Dispensation from formal ethical approval was sought at The Ethic Committee in Region Zealand and is awaiting a decision.

Adverse events Serious adverse events registration will be included in the participant diaries and the generic follow-up questionnaire. Any undesirable experience associated with the use of healthcare services or medication in a patient that may lead to discontinuation from the project or a longer term disruption in the personal intervention participation plan will be considered an adverse event, e.g., death, hospitalization, injury, impairment, serious illness requiring medication (somatic or psychiatric) or an increase in pain medication.

The project has no expected risks of adverse effects. In case of injury, all the participants have their right to seek patient compensation according to the current legislation rules.

Dissemination plan The project will be reported according to the Standards for QUality Improvement Reporting Excellence (SQUIRE) framework for reporting new knowledge about how to improve healthcare and the CONSORT extension for pilot and feasibility trials. All the results - positive, negative or undecisive - will be published in peer-reviewed scientific journals. The participants will receive a brief report with the results of their participation as standard.

Funding The project is funded by the Exercise First program grant from Region Zealand. External funding will be sought.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years old
* Completed their chronic pain treatment at the Multidisciplinary Pain Centre (MPC) at Naestved hospital
* Self-reported MVPA <150 min./ week)
* Diagnoses such as fibromyalgia or musculoskeletal pain in low back, knees, legs, neck, arms and shoulders

Exclusion Criteria:

* Referral to other specialized treatments or health services (e.g., delivered by rheumatologists, psychiatrists, physiotherapists or multidisciplinary)
* Not sufficient Danish writing and speaking proficiency allowing independent questionnaire completion and translation-free conversation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2024-04-17 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | Through study completion, on average 6 months
  Mean n recruited per month
Participant retention | After 3 months
  % mean of completed the assessments planned, post-intervention
Program adherence | After 3 months
  % mean of participation in the sessions planned, post-intervention
Patients' self-perceived relevance, timing and mode of delivery | After 3 months
  % mean of positive patients' feedback regarding the intervention's relevance, timing and mode of delivery, post-intervention
Assessment procedure acceptance | After 3 months
  % mean of positive response, post-intervention
Adverse events | After 3 months
  n, % caused discontinuation, post-intervention
Fidelity of delivery | After 3 months
  % of contents delivered as planned, post-intervention

SECONDARY OUTCOMES:
Change in MVPA time after 3 months | After 3 months
  MVPA will be measured by two accelerometers, worn for a week on the right thigh and the wrist will help to objectively assess MVPA
Change in Occupational performance and satisfaction after 3 months | After 3 months
  The Canadian Occupational Performance Measure (COPM) will help access self-evaluated performance and satisfaction with performance of meaningful everyday occupations in the areas of self-care, productivity and leisure, using a semi-structured interview and two scores - for performance and satisfaction with performance
Change in Occupational balance after 3 months | After 3 months
  Occupational Balance Questionnaire (OBQ) will evaluate the activity balance after MVPA optimization as an outcome important for healthy lifestyle maintenance
Change in Pain intensity after 3 months | After 3 months
  Pain intensity will be assessed by 0-10 VAS, min. and max. levels
Change in Pain self-efficacy after 3 months | After 3 months
  Pain Self-Efficacy questionnaire (PSEQ), a 10-item self-report measure will evaluate pain self-management regarding domestic chores, social life, productivity and need of medication (7-point Likert scales from 0 = not at all confident to 6 = completely confident)
Change in Pain spreading after 3 months | After 3 months
  Body Pain Chart representing 45 anatomic regions in anterior and posterior body positions to quantify pain spreading as an indicator for pain sensitivity
Change in Central sensitization after 3 months | After 3 months
  Central Sensitization Inventory (CSI-Dan) to evaluate central nervous system sensitivity that may have influence on PA and overall well-being
Change in Pain catastrophizing after 3 months | After 3 months
  The Pain Catastrophizing Scale (PCS), a 13-item self-report measure will assess pain-related catastrophic thinking (5-point Likert scales from 0 = not at all to 4 = all the time)
Change in Sleep quality after 3 months | After 3 months
  Karolinska Sleep Questionnaire (KSQ), a 13-item self-report measure will monitor sleep quality in the last 3 months (5-point Likert scales from 1 = never/ very good to 5 = always/ very bad)
Change in Health-related quality of life (HRQoL) after 3 months | After 3 months
  EQ-5D-5L will deliver the outcome measure comparable with previous HRQoL assessments in the chronic pain cohort and the Danish general population norms (the EQ-5D-5L Index values also include the assessment of problems related to mobility, pain/discomfort, usual activities and anxiety/ depression that will support other relevant assessments)
Change in Treatment satisfaction after 3 months | After 3 months
  Overall satisfaction with the intervention briefly assessed by a 5-point Likert scale developed for the project, from 0 = not satisfied at all to 4 = very satisfied)

OTHER OUTCOMES:
Accessibility after 3 months | After 3 months
  Individual opinions on the availability of the intervention, assessed by a semi-structured interview
Practicability after 3 months | After 3 months
  Individual opinions on the intervention as functional, suitable, or demanding additional training, assessed by a semi-structured interview
Accept after 3 months | After 3 months
  Individual opinions on whether the clients considered the intervention acceptable, assessed by a semi-structured interview

CONTACTS AND LOCATIONS:
Overall Officials: Søren T. Skou, PhD, Study Director — Department of Physiotherapy and Occupational Therapy; Lars Tang, PhD, Study Chair — Department of Physiotherapy and Occupational Therapy
Locations (1):
- Naestved, Slagelse and Ringsted Hospitals, Slagelse, Region Sjælland, Denmark